CLINICAL TRIAL: NCT04981392
Title: Trusted Messengers: Supporting Physicians in Promoting COVID-19 Vaccination
Brief Title: Trusted Messengers: Intervention to Promote COVID-19 Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Kimberly Fisher, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H00023254; 1R01MD016883-01 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Covid19; Vaccination
Keywords: Covid-19; Vaccine Hesitancy; Vaccine Confidence
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: The intervention will be tested using a pragmatic, cluster randomized clinical trial. Randomization will occur at the clinic level. Clinics will be matched by practice setting (Academic, Community, Federally Qualified Health Center) and other characteristics as possible. Within each pair, clinics will be randomly allocated to either the intervention or usual care Arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Primary care text message outreach to unvaccinated patients and resources to support PCPs
  Interventions: Behavioral: Primary care text message outreach to unvaccinated patients and resources to support PCPs
- Control Arm (No Intervention): Patients will receive usual care

INTERVENTIONS:
Behavioral: Primary care text message outreach to unvaccinated patients and resources to support PCPs — Patients: Eligible patients will receive a series of text messages from their PCP or primary care clinic recommending a study website as a trusted source of information about the COVID-19 vaccines and information on how and where to schedule a vaccination.
  Providers: PCPs will receive resources to support their conversations with patients about the COVID-19 vaccines (factsheets, prescription pads, electronic "smartphrase").
  Arms: Intervention Arm

SUMMARY:
The study aims to assess the impact of a multicomponent intervention to support Primary Care Provider (PCP) outreach to promote COVID-19 vaccination among vulnerable patients in and near Worcester, MA via a pragmatic, cluster randomized trial.

DETAILED DESCRIPTION:
The goal of this study is to increase uptake of the COVID-19 vaccine among vulnerable populations through systematic primary care (PCP or clinic) text message outreach to unvaccinated patients, information provision via a study website, and resources to support PCPs.

The clinical trial will randomize 14 primary care clinics from three health systems in the Worcester, Massachusetts area to intervention or control. Eligible patients seen at a study clinic randomized to the intervention will receive a series of text messages from their PCP or primary care clinic recommending a study website as a trusted source of information about the COVID-19 vaccines and information on how and where to schedule a vaccination.

Providers at a study clinic randomized to the intervention will be provided resources to support their conversations with unvaccinated patients during the intervention. Resources will include access to the study website, factsheets to share with vaccine hesitant patients, prescription pads to be used to "prescribe' the website, and an electronic "smartphrase" that can automatically add information about the study website and how to schedule a COVID-19 vaccination to patients' After Visit Summary and/or clinic note.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen by a PCP at a participating clinic site within 3-years prior to study start
* Age > / = 18 years

Exclusion Criteria:

* Patients who have received at least one dose of a COVID-19 vaccine series prior to the start of the intervention
* Non-Massachusetts residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21844 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Fisher, M.D, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 primary care clinics from three health systems in Central Massachusetts - a tertiary care academic medical center with community practices and two local Federally Qualified Health Centers were included in the study. The 14 participating clinics were matched according to size, practice setting (academic, community, FQHC), availability of COVID-19 vaccines in-clinic, and baseline COVID-19 vaccination rates and block randomized in 4 blocks.
Pre-assignment Details: Eligible participants included patients seen at one of the study clinics within 3-years period prior to start of the intervention, age >= 18 years, who had not been vaccinated against COVID-19 and were Massachusetts residents.
Units Other Than Participants: Clinic Sites
Groups:
- Intervention Arm: Primary care text message outreach to unvaccinated patients and resources to support PCPs
  Primary care text message outreach to unvaccinated patients and resources to support PCPs: Patients: Eligible patients will receive a series of text messages from their PCP or primary care clinic recommending a study website as a trusted source of information about the COVID-19 vaccines and information on how and where to schedule a vaccination.
  Providers: PCPs will receive resources to support their conversations with patients about the COVID-19 vaccines (factsheets, prescription pads, electronic "smartphrase").
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 10996; 7 Clinic Sites | 10848; 7 Clinic Sites
Completed | 10996; 7 Clinic Sites | 10848; 7 Clinic Sites
Not Completed | 0; 0 Clinic Sites | 0; 0 Clinic Sites

BASELINE CHARACTERISTICS:
Population: Patients that are ≥18, unvaccinated, visit at study clinic in past 3 years, alive at time of data pull, MA residents.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 10,996 | 10,848 | 21844
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 79 | 140 | 219
  Between 18 and 65 years | 9649 | 9720 | 19369
  >=65 years | 1268 | 988 | 2256
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 6156 | 6134 | 12290
  Male | 4839 | 4714 | 9553
  Unknown/Missing | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3937 | 4466 | 8403
  Not Hispanic or Latino | 6676 | 6171 | 12847
  Unknown or Not Reported | 383 | 211 | 594
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 66 | 31 | 97
  Asian | 314 | 153 | 467
  Native Hawaiian or Other Pacific Islander | 76 | 53 | 129
  Black or African American | 1462 | 705 | 2167
  White | 5913 | 6032 | 11945
  More than one race | 875 | 2889 | 3764
  Unknown or Not Reported | 2290 | 985 | 3275
Region of Enrollment [Number; unit: participants]
  United States | 10996 | 10848 | 21844

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Vaccination Within 3 Months
Description: The number of patients in the intervention and control arms who receive at least one dose of a COVID-19 vaccination within 3 months of the last text message being sent will be ascertained via the Electronic Health Record (EHR).
Time Frame: 3 months
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 10996 | 10848
Participants | 137 | 98
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Test type: Superiority; p = 0.0066, Difference in adjusted % vaccinated; Cox Proportional Hazard = 0.49, Standard Error of Mean 0.18

2. Secondary Outcome: COVID-19 Vaccination Within 6 Months
Description: The number of patients in the intervention and control arms who receive at least one dose of a COVID-19 vaccination within 6 months of the last text message being sent will be ascertained via the Electronic Health Record (EHR).
Time Frame: 6 months
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 10996 | 10848
Participants | 235 | 162
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Test type: Superiority; p = 0.0058, Difference in adjusted % vaccinated; Cox Proportional Hazard = 0.83, Standard Error of Mean 0.30

ADVERSE EVENTS:
Time Frame: Deaths and Adverse Events were not collected
Description: Deaths and Adverse Events were not collected
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT04981392/Prot_SAP_000.pdf